CLINICAL TRIAL: NCT02691923
Title: Diagnostic Performance of Fluorescein as an Intraoperative Brain Tumor Biomarker: Correlation With Preoperative MR, ALA-induced PpIX Fluorescence, and Histopathology
Brief Title: Diagnostic Performance of Fluorescein as an Intraoperative Brain Tumor Biomarker
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: David W. Roberts (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David W. Roberts, Professor of Surgery (Neurosurgery), Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: D12090; R01NS052274-01A2 (NIH)
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Brain Cancer
Keywords: High Grade Glioma; Low Grade Glioma; Brain Tumor
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Fluorescein; Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Fluorescein (Active Comparator): Fluorescein administered IV at 5mg/kg approximately 30 minutes prior to the beginning of the tumor resection. A second injection may occur if the fluorescein fluorescence is dissipated substantially during the course of the procedure.
  Interventions: Drug: Fluorescein
- Fluorescein + ALA (Experimental): Fluorescein administered IV at 5mg/kg approximately 30 minutes prior to the beginning of the tumor resection. A second injection may occur if the fluorescein fluorescence is dissipated substantially during the course of the procedure.
  ALA administered orally at 20mg/kg approximately 3 hours before surgery.
  Interventions: Drug: Fluorescein + ALA

INTERVENTIONS:
Drug: Fluorescein
  Other Names: Fluorescite
  Arms: Fluorescein
Drug: Fluorescein + ALA
  Other Names: Flourescein = Fluorescite; ALA = 5-Aminolevulinic Acid
  Arms: Fluorescein + ALA

SUMMARY:
This clinical research will evaluate the diagnostic potential of fluorescein as visualized through an operating microscope relative to 1) contrast enhancement on co-registered preoperative MR scans, 2) intraoperative ALA-induced PpIX fluorescence and 3) gold-standard histology obtained from biopsy sampling during the procedure.

Subjects will include those people with operable brain tumor with first-time presumed pre-surgical diagnosis of high-grade glioma or low-grade glioma.

DETAILED DESCRIPTION:
Consenting subjects who have met inclusion and exclusion criteria will be enrolled to receive either fluorescein+ALA or fluorescein alone. HGG patients will be randomized on a 2 to 1 basis to receive either both fluorescein and ALA or fluorescein alone, and LGG patients will be randomized on a 1 to 1 basis.

This study is a diagnostic trial of fluorescein fluorescence as an intraoperative imaging biomarker during open cranial surgery for tumor resection of first-time (preoperatively) presumed high or low grade glioma. Subjects participate in a "one-time" event/visit (i.e, surgery) as part of this protocol. Images and data from the patient's pre- and post-operative MR scans are used for analysis in the study, but these acquisitions are part of the patient's standard-of-care, would occur independently of whether the participant is enrolled; and thus, are not considered to be research study visits. No post-surgical follow-up visit is part of the protocol data collection or analysis. Patients are monitored for possible adverse events through the routine follow-up under the care of the operating surgeon involved in the study procedures, post-operatively and subsequently through the medical record. Hence, this information is already being collected as part of standard-of-care and is available for adverse event surveillance. Patients receiving ALA who present with abnormally elevated LFTs beyond the peri-operative observation period are monitored on a regular basis until resolution and this blood testing is considered to be part of the study.

Administration of study drug:

Patients enrolled in the fluorescein+ALA arm will be administered orally 5-ALA (DUSA Pharmaceuticals, Tarrytown, NY) at 20 mg/kg body weight, dissolved in 100 ml of water, approximately 3 hours prior to the induction of anesthesia.

For patients receiving only fluorescein, the operating surgeon will request bolus injection (at a dose of 5 mg/kg) approximately 30 minutes prior to the start of tumor resection. For especially long cases (e.g., > 4 h) or if fluorescein fluorescence dissipates substantially during the course of the procedure, a second bolus injection may occur later in the case.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative diagnosis of either presumed first-time low or high grade glioma (astrocytoma, oligodendroglioma, mixed oligo-astrocytoma, anaplastic astrocytoma, and glioblastoma multiforme).
2. Tumor judged to be suitable for open cranial resection based on preoperative imaging studies.
3. Valid informed consent by subject or subject's LAR.
4. No serious associated psychiatric illnesses.
5. Age ≥ 21 years old.

Exclusion Criteria:

1. Pregnant women or women who are breast feeding.
2. History of hypersensitivity to fluorescein.
3. History of cutaneous photosensitivity, porphyria, hypersensitivity to porphyrins, photodermatosis, exfoliative dermatitis.
4. History of liver disease within the last 12 months.
5. Elevated LFTs (AST, ALT, ALP or bilirubin levels greater than 2.5 times the normal limit) from laboratory tests conducted within 30 days prior to surgery.
6. Serum creatinine in excess of 180µmol/L (2.04 md/dL) within 30 days prior to surgery.
7. Inability to comply with the photosensitivity precautions associated with the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fluorescein performance as an intraoperative biomarker for tumor tissue will be reported. | 24 months
  The predictive performance of fluorescein fluorescence as an intraoperative imaging biomarker of tumor during surgery in patients with a clinical diagnosis of high grade glioma (HGG) and patients with a clinical diagnosis of low grade glioma (LGG) will be measured. Fluorescence will be measured both quantitatively via an intraoperative probe and visually by the neurosurgeon through the operating microscope. Endpoints will be assessed separately for HGG and LGG groups.

SECONDARY OUTCOMES:
Fluorescein performance as visualized and measured with an intraoperative probe will be reported | 24 months
  The performance of fluorescein as visualized by the neurosurgeon and measured quantitatively with an intraoperative probe will be analyzed to the contrast-enhancement on coregistered preoperative MR scans in patients with a clinical diagnosis of high grade glioma.
Fluorescein versus fluorescein + ALA performance will be reported in patients in patients with 2 different types of tumors | 24 months
  The performance of fluorescein versus fluorescein + ALA as visualized by the neurosurgeon and measured quantitatively with an intra-operative probe will be analyzed in patients with a clinical diagnosis of either high grade glioma (HGG) or low grade glioma (LGG).

CONTACTS AND LOCATIONS:
Overall Officials: David W Roberts, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Sally B Mansur, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roberts DW, Valdes PA, Harris BT, Hartov A, Fan X, Ji S, Leblond F, Tosteson TD, Wilson BC, Paulsen KD. Glioblastoma multiforme treatment with clinical trials for surgical resection (aminolevulinic acid). Neurosurg Clin N Am. 2012 Jul;23(3):371-7. doi: 10.1016/j.nec.2012.04.001. PMID 22748650
- [Background] Elliott JT, Dsouza AV, Davis SC, Olson JD, Paulsen KD, Roberts DW, Pogue BW. Review of fluorescence guided surgery visualization and overlay techniques. Biomed Opt Express. 2015 Sep 3;6(10):3765-82. doi: 10.1364/BOE.6.003765. eCollection 2015 Oct 1. PMID 26504628
- [Background] Valdes PA, Jacobs V, Harris BT, Wilson BC, Leblond F, Paulsen KD, Roberts DW. Quantitative fluorescence using 5-aminolevulinic acid-induced protoporphyrin IX biomarker as a surgical adjunct in low-grade glioma surgery. J Neurosurg. 2015 Sep;123(3):771-80. doi: 10.3171/2014.12.JNS14391. Epub 2015 Jul 3. PMID 26140489